CLINICAL TRIAL: NCT03886714
Title: Screening for Fabry Disease in Renal Transplantation
Acronym: DEFYT
Status: Terminated | Type: Observational
Why Stopped: Low recreuitement numbers and end of grant.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0015; UF 7561 (Other: Montpellier University Hospital)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease; Nephropathy
Keywords: Fabry disease; Renal transplantation; Diabetic nephropathy; Focal Segmental Hyalinosis (FSH); Undetermined nephropathy
MeSH Terms: conditions — Fabry Disease; Kidney Diseases; Diabetic Nephropathies | interventions — Mass Screening; Early Detection of Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 9 mL EDTA (ethylenediaminetetraacetic acid) blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening for Fabry disease — Screening for the α-galactosidase (GAL) enzyme activity (men + women) and plasma Lyso globotriaosylsphingosine (GL3, women) for the diagnosis of Fabry disease.
Diagnostic Test: Screen for α-galactosidase mutation — If necessary (positive for GAL), genetic confirmation tests for Fabry disease will be performed (men + women).

SUMMARY:
Single centre, prospective pilot study examining the relevance to screen for Fabry disease in a cohort of patients who have undergone renal transplantation for nephropathy of indeterminate cause, vascular nephropathy, diabetic nephropathy or secondary focal segmental hyalinosis with no established cause.

DETAILED DESCRIPTION:
Exploration whether Fabry disease cases can be identified among patients who are followed at the Montpellier University Hospital after renal transplantation, with indeterminate cause of renal failure or diabetic nephropathy (due to its high frequency) or secondary focal segmental hyalinosis (FSH).

At the population level, the identification of cases at the Montpellier centre could then justify to expand this screening to other French centres. The goal is to contribute to adapt current guidelines of renal failure assessment, by systematically including Fabry among the diagnostic tests. Whether all patients with renal failure are concerned, or only those with indeterminate cause, is an important question this study will address.

ELIGIBILITY:
Inclusion Criteria:

* Nephropathy of indeterminate cause, or secondary FSH or diabetic nephropathy
* Patients with kidney transplanted
* Patients still followed at the Montpellier University Hospital
* Obtaining written informed consent
* Age > 18 years old, no upper age limit

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified from a database, who have undergone renal transplantation for nephropathy of indeterminate cause, vascular nephropathy, diabetic nephropathy or secondary focal segmental hyalinosis with no established cause, and still followed at the Montpellier University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Positive screen result | Inclusion visit
  The genetic analysis will be performed based on the biochemical results (low enzyme activity, raised lysoGL3)

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No